CLINICAL TRIAL: NCT02683408
Title: Diosmiplex (Vasculera®) in Primary and Secondary Raynaud's Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PVR-02
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Raynaud's Disease
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- diosmiplex (Experimental): diosmiplex 630 mg BID administered orally
  Interventions: Dietary Supplement: diosmiplex
- placebo (Placebo Comparator): placebo BID administrered orally
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — inactive placebo
  Arms: placebo
Dietary Supplement: diosmiplex — diosmiplex is an FDA regulated medical food product
  Other Names: Vasculera
  Arms: diosmiplex

SUMMARY:
Diosmiplex is a product marketed for the management of diseases due to venous and microvascular dysfunction. Raynaud's phenomenon is a disorder of characterized by spasm of small arteries and impaired microvascular flow. This study will examine the effects of diosmiplex on the frequency and severity of Raynaud's episodes in susceptible people.

DETAILED DESCRIPTION:
Raynaud's phenomenon is a disorder characterized by spasm of digital arteries leading to blanching, coldness and discomfort of the affected digit, affecting up to 3-5% of the population at some time in their lives. Raynaud's is roughly classified into primary and secondary forms. The primary form may occur without apparent cause or following such things as acute trauma, repetitive vibrating trauma or frostbite. Secondary Raynaud's occurs in association with a variety of systemic immunological diseases such as rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), systemic sclerosis (SS) and Sjogren's syndrome. Perhaps the most severe forms are associated with systemic sclerosis, less often in SLE where severe microvascular changes can lead to digital ulcerations which are difficult to heal and produce considerable functional impairment Treatment of Raynaud's has been a significant clinical challenge. The primary modality is to avoid cold exposure. Many drug classes have been shown to have some, but highly variable and potential toxicities.

Diosmiplex is a prescription medical food product composed of the botanical based flavonoid molecule, diosmin, and a proprietary systemic blood alkalinizing agent, Alka4-complex. Diosmin has been used successfully in Europe as a drug for chronic venous insufficiency and its complications, including venous ulcers for more than 35 years. There is a large body of published literature regarding the molecular activity, clinical efficacy and safety of the active molecule in diosmin as well as its effects on the microvasculature where it has been shown to reduce inflammation, improve structural integrity, reduce capillary damage and improve capillary flow but no prospective clinical studies have been published regarding its effect in Raynaud's phenomenon. This will be the first prospective study to examine the efficacy and safety of diosmin, as diosmiplex, in both primary and secondary Raynaud's. The study will intentionally seek to enroll a subset of subjects with scleroderma with Raynaud's complicated by digital ulcers.

This will be a two (2) month randomized, double blind, placebo controlled study. Patients with either primary or secondary Raynaud's phenomenon present for at least 12 months and either untreated or inadequately controlled on therapy, defined as having at least four (4) vasospastic episodes/week, will be eligible for enrollment

ELIGIBILITY:
Inclusion Criteria:

* either gender, ages 18-80
* established diagnosis of primary or secondary Raynaud's phenomenon
* minimum of 4 vasospastic episodes/week
* medication specifically for Raynaud's must be stable for 30 days prior to the screening visit and must be maintained unchanged for the duration of the study medication specifically for digital ulceration must be stable for 60 days prior to the screening visit and must be maintained unchanged for the duration of the study
* not pregnant or breast feeding
* using approved method of birth control if capable of becoming pregnant (Appendix II)
* capable of reading and understanding the informed consent document

Exclusion Criteria:

* pregnant or nursing women
* any change in dose of oral medication specifically for Raynaud's or digital ulcers including, but not limited to, vasodilators, adrenergic blockers, antihypertensives, calcium channel blockers, ACE inhibitors, phosphodiesterase inhibitors (e.g., sildenofil,) endothelin receptor antagonists (e.g., bosentan), prostanoids (e.g., iloprost) within the 30 days prior to the screening visit for Raynaud's and /or 60 days for digital ulcers and during the duration of the study.
* any intravenous or intra-arterial Raynaud's therapy within 1 month prior to the screening visit
* Raynaud's secondary to mechanical (non-thermal) trauma
* concomitant use of diclofenac or metronidazole
* history of unstable coronary artery disease, chronic hepatic disease with ALT, AST, or alkaline phosphatase >1.3 time upper limit of normal for reference laboratory, renal disease with serum creatinine >2.5 or any gastrointestinal disease that could potentially interfere with absorption of the study product.
* history of substance abuse including "recreational drugs" and/or alcohol intake in excess of one unit daily. For the purposes of this study a unit of alcohol is defined as 12 ox. of beer, 6 oz. of wine or 1.5 oz. of hard liquor.
* history of any significant medical condition that, in the opinion of the investigator might put the subject at risk in this trial
* participation in another clinical trial within 30 days of the screening visit or 7 half lives of the study product, whichever is longer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
percentage of subjects with by at least 50% reduction in number of vasospastic episodes | 8 weeks
  For each primary and secondary endpoint, the number and percentage of subjects meeting the criterion will be presented by treatment group at Week 4 and Week 8.

SECONDARY OUTCOMES:
percentage of subjects with at least 50% reduction in severity of vasospastic episodes | 8 eeks
  For each primary and secondary endpoint, the number and percentage of subjects meeting the criterion will be presented by treatment group at Week 4 and Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Levy, MD, Study Director — Primus Pharmaceuticals
Locations (11):
- United States (11):
  - Sun Valley Arthritis Center, Peoria, Arizona
  - Advanced Arthritis Care and Research, Scottsdale, Arizona
  - Valerius Medical Group, Los Alamitos, California
  - Science and Research Institute, Inc., Jupiter, Florida
  - Jeffrey Alper, MD, Naples, Florida
  - Steven Kimmel MD, Tamarac, Florida
  - Diagnostic Rheumatology, Indianapolis, Indiana
  - Arthritis Treatment Center, Frederick, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - West Virginai Research Institute, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No